CLINICAL TRIAL: NCT04326998
Title: Natural Gutta-percha Solvent Did Not Affect Postoperative Pain in Retreatment: a Randomized Clinical Trial
Brief Title: Gutta-percha Solvent on Postoperative Pain After Root Canal Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2019/054.2608
Record Dates: First submitted 2020-03-27; First posted 2020-03-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Root Canal; Retreatment
MeSH Terms: conditions — Pain, Postoperative | interventions — Solvents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-solvent (Active Comparator): mechanical or heat treatment
  Interventions: Procedure: non-solvent
- solvent (Experimental): GuttaClear
  Interventions: Procedure: solvent

INTERVENTIONS:
Procedure: solvent — using solvent (GuttaClear) in procedure
  Arms: solvent
Procedure: non-solvent — non-solvent
  Arms: non-solvent

SUMMARY:
The process of non-surgical retreatment includes removing the previous root canal filling materials, disinfecting and sealing the root canal system to prevent re-infection. Gutta-percha is the most common root canal filling material used with various types of sealers. To remove gutta-percha, solvent has been suggested because of its ability to dissolve gutta-percha. The new formula, under the brand name, GuttaClear, has been investigated for its comparable dissolving ability and lower cytotoxicity when compared with others that are currently used. However, no information is currently available of GuttaClear solvent concerning postoperative pain. Therefore, the present study will evaluate postoperative pain after non-surgical retreatment cases using GuttaClear as a solvent compared with no solvent used. Sixty participants are chosen and distributed into 2 groups, randomly. After the procedures, participants will receive the questionnaires about postoperative pain and the amount of medication intake. Both will be recorded at six time periods: (1) immediately after procedure; (2) 6 hours after procedure; (3) 12 hours after procedure; (4) 24 hours after procedure; (5) 48 hours after procedure and (6) 72 hours after procedure.

ELIGIBILITY:
Inclusion Criteria:

* not be contra-indicated with medication used in this study (ibuprofen)
* have a previously treated endodontic single-root tooth with the need of retreatment
* all those teeth must be restorable
* old root canal filling materials must be located at 1 to 3 mm from the radiographic apex in the periapical radiograph

Exclusion Criteria:

* open apex, root resorption or root perforation
* participants presenting pre-operative pain and/or swelling at the appointment visit
* taking analgesics or antibiotics less than one week before appointment visit
* experiencing problems in completing the pain questionnaires
* tooth which does not contain gutta-percha
* cannot be patent through the apex at the appointment visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 3 days
  NRS score recorded from 0 to 10 while 0 means no pain and 10 means the worst possible pain

SECONDARY OUTCOMES:
number of Ibuprofen intake | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Duangrat Sirijindamai, DDS, Principal Investigator — Mahidol University
Locations (1):
- Mahidoluniversity, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jantarat J, Malhotra W, Sutimuntanakul S. Efficacy of grapefruit, tangerine, lime, and lemon oils as solvents for softening gutta-percha in root canal retreatment procedures. J Investig Clin Dent. 2013 Feb;4(1):60-3. doi: 10.1111/j.2041-1626.2012.00143.x. PMID 23382062
- [Result] Genc Sen O, Erdemir A, Canakci BC. Effect of solvent use on postoperative pain in root canal retreatment: a randomized, controlled clinical trial. Clin Oral Investig. 2020 Jan;24(1):257-263. doi: 10.1007/s00784-019-02948-3. Epub 2019 May 15. PMID 31093742
- [Result] Topcuoglu HS, Topcuoglu G. Postoperative pain after the removal of root canal filling material using different techniques in teeth with failed root canal therapy: a randomized clinical trial. Acta Odontol Scand. 2017 May;75(4):249-254. doi: 10.1080/00016357.2017.1283707. Epub 2017 Feb 5. PMID 28162017
- [Result] Garcia-Font M, Duran-Sindreu F, Morello S, Irazusta S, Abella F, Roig M, Olivieri JG. Postoperative pain after removal of gutta-percha from root canals in endodontic retreatment using rotary or reciprocating instruments: a prospective clinical study. Clin Oral Investig. 2018 Sep;22(7):2623-2631. doi: 10.1007/s00784-018-2361-x. Epub 2018 Feb 2. PMID 29396645
- [Derived] Sirijindamai D, Wichai W, Mitrirattanakul S, Jantarat J. Effect of GuttaClear on Postoperative Pain After Root Canal Retreatment: A Randomized Clinical Trial. Eur Endod J. 2023 Jan;8(1):55-64. doi: 10.14744/eej.2022.85047. PMID 36748447